CLINICAL TRIAL: NCT03654963
Title: Parallel Group Randomized Controlled Trial to Assess the Impact of Medication Reconciliation at Hospital Admission on Healthcare Outcomes
Brief Title: Study to Assess the Impact of Medication Reconciliation at Hospital Admission on Healthcare Outcomes
Acronym: MedRec
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Alessandro Ceschi, Medical and scientific director of the Istituto di Scienze Farmacologiche della Svizzera Italiana, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Safety Issues
Keywords: medication reconciliation; safe pharmacotherapy
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Intervention Model Description: Allocation: centralized randomization; a unique list of randomization will be generated by the clinical trial unit (CTU) of the EOC with an ad hoc software, and patients will be allocated 1:1 in either the intervention or the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only pharmacy assistants and clinical pharmacists, who will obtain the best possible medication history and perform medication reconciliation, will know the assignment to either the intervention or the control group. Participants and outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients of the control group will not receive the best possible medication history with medication reconciliation at admission. The standard physician-acquired medication history will be performed as usual.
- Medication reconciliation (Experimental): The pharmacy assistant will obtain the best possible medication history by compiling a comprehensive list of the medications the patient is taking. To confirm the accuracy of the history, the pharmacy assistant will use at least two sources of information, one of which being, when possible, the interview with the patient and/or family members. The clinical pharmacist will reconcile the best possible medication history with prescribed medicines and, to resolve unclear or ambiguous discrepancies between the two lists and/or to propose any adaptations of the pharmacotherapy, the clinical pharmacist will refer to the medical doctor. The medical doctor will decide potential changes in pharmacotherapy and communicate them to the patient.
  Interventions: Procedure: Medication reconciliation

INTERVENTIONS:
Procedure: Medication reconciliation — Medication reconciliation is the systematic process described above.
  Arms: Medication reconciliation

SUMMARY:
Medication reconciliation is a systematic process by which health care professionals obtain the most complete and accurate information about the drugs regularly taken by patients. Internationally, the value of this procedure is mainly attributed to the reduction in the number of adverse drug events, which can cause drug-related morbidity and mortality, as well as unnecessary health care costs.

As part of the Progress! Pilot project Safe Pharmacotherapy at the interface points, promoted by the Federal Office of Public Health, coordinated by the Swiss Patients Safety Foundation and held in several Swiss hospitals, medication reconciliation at hospital admission was introduced at the regional hospital Beata Vergine in Mendrisio, from 2014 to 2016. During this pilot project it was shown that medication reconciliation after obtaining the best possible medication history by a pharmacist at hospital admission, in comparison with the standard medication history obtained by the physician at admission, reduced the number of clinically relevant drug discrepancies.

A structured, well-established and practicable procedure of medication reconciliation that improves patient safety assuring a better quality of care at hospital admission might provide evidence that medication reconciliation could be a valuable intervention to be applied systematically in all EOC hospitals at admission, as well as subsequently potentially at the other hospital interfaces.

The purpose of this study is to evaluate whether obtaining the best possible medication history and performing medication reconciliation at hospital admission results in improving some specific healthcare outcomes.

The study seeks primarily to determine if obtaining the best possible medication history and performing medication reconciliation, in comparison with the standard medication history, reduces the number of subsequent unplanned all-cause hospital visits (readmissions and emergency department visits within 30 days after initial discharge). As secondary objectives, the study aims at assessing if best possible medication history with medication reconciliation, in comparison with the standard medication history, reduces the incidence of adverse drug reactions during hospital stay, shortens length of stay, leads to a reduction in the use of hospital resources, and/or is associated with a decreased number of deaths.

DETAILED DESCRIPTION:
Patients of the control group will not receive the best possible medication history with medication reconciliation at admission. The standard physician-acquired medication history will be performed as usual.

Eligible patients, randomized within the intervention arm, will receive medication reconciliation according to the following steps:

1. The pharmacy assistant will obtain the best possible medication history by compiling a comprehensive list of the medications the patient is taking and details about how the drugs are taken. In order to confirm the accuracy of the history, the pharmacy assistant will use at least two sources of information, one of which being, when possible, the interview with the patient and/or family members, in addition to referral letters, prescriptions and drug lists from primary care centres, and other.
2. The clinical pharmacist will reconcile best possible medication history with prescribed medicines and, to resolve unclear or ambiguous discrepancies between the two lists and/or to propose any adaptations of the pharmacotherapy, the clinical pharmacist will refer to the medical doctor.
3. The medical doctor will decide potential changes in pharmacotherapy and communicate them to the patient providing complete information on medicines.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the inpatient wards of the two regional hospitals Beata Vergine in Mendrisio and La Carità in Locarno, fulfilling one of the following inclusion criteria, will be eligible for the study:

* patients aged ≥ 85 years
* patients with > 10 drugs at admission

Patients with home care as well as patients from elderly homes, meeting the inclusion criteria, will be factored in the study population.

Eligible patients will be included one-time only.

Exclusion Criteria:

The presence of any of the following exclusion criteria will lead to patient exclusion:

* patients admitted to intensive care unit who do not reach inpatient wards
* patients who are planned to stay within inpatient wards for less than 48 hours
* patients who have been admitted to any of the EOC hospital wards within the previous 3 months and have been discharged at home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1702 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Composite post-discharge healthcare use variable | Within 30 days after initial discharge
  Total number of unplanned all-cause hospital visits (readmissions and emergency department visits within 30 days after initial discharge).

SECONDARY OUTCOMES:
Incidence of ADRs during hospital stay | 1 year
  To measure the incidence of ADRs developed by patients during the hospital stay, the active pharmacovigilance system currently in use at the Centro Regionale di Farmacovigilanza del Canton Ticino, will be exploited. EMRs identified through this system and referring to patients from both the two study sites, aged ≥85 years or with more than 10 medications at admission, will be manually validated (to discard false positive cases). Subsequently, ADRs will be categorized as not serious or serious (according to the WHO seriousness criteria, for resulting in death, being life threatening, prolonging hospitalization, resulting in persistent disability or incapacity and other). Outcome assessor will be masked to group allocation. At the end of the analysis, ADRs will be matched to either the intervention or the control group
Length of hospital stay | 1 year
Death during hospital stay | 1 year
Number of resources used during hospital stay | 1 year
  Laboratory tests, radiologic exams, echocardiography, electrocardiograms

CONTACTS AND LOCATIONS:
Overall Officials: Dr med Alessandro Ceschi, PD, FEAPCCT, Principal Investigator — Institute of Pharmacological Science of Southern Switzerland, Ente Ospedaliero Cantonale
Locations (2):
- Switzerland (2):
  - Regional Hospital La Carità, Locarno
  - Regional Hospital Beata Vergine, Mendrisio

REFERENCES:
- [Derived] Ceschi A, Noseda R, Pironi M, Lazzeri N, Eberhardt-Gianella O, Imelli S, Ghidossi S, Bruni S, Pagnamenta A, Ferrari P. Effect of Medication Reconciliation at Hospital Admission on 30-Day Returns to Hospital: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2124672. doi: 10.1001/jamanetworkopen.2021.24672. PMID 34529065